CLINICAL TRIAL: NCT05992220
Title: A Randomized, Multicenter, Open-Label, Phase II Trial of Atezolizumab Plus Bevacizumab Alone or Combined with External Beam RadioTherapy for HepatoCellular Carcinoma with Macrovascular Invasion (ALERT-HCC)
Brief Title: Atezolizumab Plus Bevacizumab Alone or Combined with External Beam Radiotherapy for HCC with Macrovascular Invasion
Acronym: ALERT-HCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Seoul National University Hospital (Other); Hanyang University Guri Hospital (Other); Soon Chun Hyang University (Other)
Responsible Party: Principal Investigator, Ju Hyun Shim, Principal Investigator, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KCT0007365; KCT0007365 (Registry Identifier: CRIS (International Clinical Trials Registry Platform))
Record Dates: First submitted 2023-07-27; First posted 2023-08-15 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-01

CONDITIONS: Hepatocellular Carcinoma; Hepatocellular Cancer; Hepatocellular Carcinoma Non-resectable; Hepatocellular Carcinoma Stage IV; Liver Cancer
Keywords: HCC; vascular invasion; portal vein tumor thrombosis; BCLC stage C
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Intervention Model Description: randomized, multicenter, open-label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Radiotherapy combination (Experimental): Atezolizumab+Bevacizumab, combined EBRT to vascular invasion
  * Atezolizumab will be administered by IV, 1200 mg on day 1 of each 21day cycle.
  * Bevacizumab will be administered by IV, 15 mg/kg on day 1 of each 21day cycle.
  * The external beam radiotherapy will commence after day 2 of the first cycle of A+B, and will be delivered in accordance with institutional protocol.
  Interventions: Radiation: Atezolizumab plus bevacizumab, combined EBRT to vascular invasion
- Atezolizumab+Bevacizumab (Active Comparator): * Atezolizumab will be administered by IV, 1200 mg on day 1 of each 21day cycle.
  * Bevacizumab will be administered by IV, 15 mg/kg on day 1 of each 21day cycle.
  Interventions: Drug: Atezolizumab plus bevacizumab

INTERVENTIONS:
Radiation: Atezolizumab plus bevacizumab, combined EBRT to vascular invasion — The external beam radiotherapy will commence after day 2 of the first cycle of atezolizumab+bevacizumab, and will be delivered in accordance with institutional protocol.
  3D-conformal radiotherapy technique is used to determine target volumes, radiation ports, and dose prescriptions by using a 3D radiotherapy planning system.
  The gross tumor volume (GTV) includes vascular invasion and a 2-cm margin into the contiguous HCC. The GTV can consist of the entire HCC and vascular invasion at the discretion of the investigator.
  The target dose is 45 Gy, however, the total dose can be reduced as low as 30 Gy according to the liver function, liver volumes, or the maximum dose to the stomach/duodenum during the planning process according to the judgment of the radiation oncologist of each participating sites.
  Arms: Radiotherapy combination
Drug: Atezolizumab plus bevacizumab — Atezolizumab plus bevacizumab q3w
  Arms: Atezolizumab+Bevacizumab

SUMMARY:
The recent global IMbrave150 study evaluated the combination of atezolizumab and bevacizumab versus sorafenib in 501 patients with advanced or metastatic Hepatocellular Carcinoma (HCC). The median overall survival (OS) was notably better in the atezolizumab/bevacizumab group. However, for HCC patients with intrahepatic macrovascular invasion (MVI), the prognosis remains poor, indicating a significant unmet need in this group.

External Beam Radiotherapy (EBRT) has shown promising results in treating HCC with MVI, especially when used in combination with trans-arterial chemoembolization (TACE). It has been reported that radiotherapy may make tumor cells more susceptible to immune-mediated therapy, potentially enhancing the effects of atezolizumab and bevacizumab.

Thus, this study aims to investigate the efficacy and safety of atezolizumab/bevacizumab alone versus atezolizumab/bevacizumab in combination with EBRT in HCC patients with macrovascular invasion.

DETAILED DESCRIPTION:
A total of 138 subjects are randomly assigned to one of two treatment groups (69 patients in the atezolizumab+bevacizumab group and 69 patients in the Atezolizumab plus Bevacizumab combined EBRT group).

* Radiotherapy combination:

  * Atezolizumab will be administered by IV, 1200 mg on day 1 of each 21day cycle.
  * Bevacizumab will be administered by IV, 15 mg/kg on day 1 of each 21day cycle.
  * The external beam radiotherapy will commence after day 2 of the first cycle of Atezolizumab+Bevacizumab, and will be delivered in accordance with institutional protocol.
* Atezolizumab+Bevacizumab:

  * Atezolizumab will be administered by IV, 1200 mg on day 1 of each 21day cycle.
  * Bevacizumab will be administered by IV, 15 mg/kg on day 1 of each 21day cycle.

Additional study identifiers: This study was also registered on the WHO's International Clinical Trials Registry Platform, CRIS, before the first participant was enrolled (ID: KCT0007365, Date of registration: 2022-06-08).

ELIGIBILITY:
Inclusion Criteria:

* Older than 19 years of age, lower than 80 years of age
* Child-Pugh class A hepatic function
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-1
* Patients with HCC [diagnosed according to AASLD guidelines] invading the intrahepatic vascular system
* No prior systemic therapy for HCC
* At least one measurable HCC lesion with ≥ 1cm diameter
* Adequate hematologic and organ function

  * Hemoglobin ≥ 9.0 g/dL
  * Absolute neutrophil count ≥ 1,000 /mm3
  * Platelet ≥ 50,000/ mm3 without transfusion
* Total bilirubin ≤ 2.5 mg/dL

Exclusion Criteria:

* Treatment history of prior systemic treatment of HCC
* Liver transplant recipients
* Patients with peptic ulcer, untreated or incompletely treated varices with bleeding or high-risk for bleeding
* Any serious illness (e.g., active infection or inflammatory condition) or uncontrolled severe medical comorbidity
* A history of treated malignancy (other than HCC) is allowable if the patient's malignancy has been in complete remission, off chemotherapy and without additional surgical intervention, during the preceding two years
* Abdominal/pelvic radiotherapy within 28 days prior to initiation of study treatment, except palliative radiotherapy to bone lesions within 7 days prior to initiation of study treatment

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2022-10-22 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
progression-free survival rate | up to approximately 3 years
  Randomization to the first occurrence of disease progression or death from any cause, whichever occurs first

SECONDARY OUTCOMES:
Overall survival rate | up to approximately 3 years
  Randomization to death from any cause, through the end of study
Objective response | up to approximately 3 years
  complete response or partial response as determined by the Investigator according to RECIST V1.1
Adverse reaction rate | through study completion, up to approximately 3 years
  Adverse reaction rate assessed by CTCAE version 5
Time to deterioration | through study completion, up to approximately 3 years
  The time from randomization to first deterioration (decrease from baseline of ≥10 points) in the patient-reported global health status (GHS) / Quality of life (QoL), physical function, or role function scales of the EORTC QLQ-C30, maintained for two consecutive assessments, or one assessment followed by death from any cause within 3 weeks
Duration of response | up to approximately 3 years
  the time interval from the date of first occurrence of a documented objective response (CR or PR, whichever status is recorded first) until the first date that disease progression or death is documented, whichever occurs first. DOR will be assessed in patients who had an objective response.
Tumor marker response (AFP, PIVKA-II) | through study completion, up to approximately 3 years
  The decrease of >20% in serum concentration of each marker from baseline across all time points during study period.

CONTACTS AND LOCATIONS:
Overall Officials: Ju Hyun Shim, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No